CLINICAL TRIAL: NCT04868383
Title: Using Smart Phone Technology to Support PrEP Uptake and Adherence in Virginia - Pilot Study
Brief Title: Using Smart Phone Technology to Support PrEP Uptake and Adherence
Acronym: prep'd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Virginia Department of Health (Other Government)
Responsible Party: Principal Investigator, Karen Ingersoll, Clinical Psychologist, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20478
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: HIV Prevention; PrEP; Adherence, Medication
Keywords: HIV; Prevention; Adherence; Uptake
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single pilot arm (Experimental): In this single arm pilot study, all participants will receive access to a novel smartphone app designed to support PrEP uptake and adherence for a 6 month period.
  Interventions: Behavioral: Use of smart phone technology to support medication adherence and uptake

INTERVENTIONS:
Behavioral: Use of smart phone technology to support medication adherence and uptake — Use of smart phone technology to support medication adherence and uptake

SUMMARY:
This is a single arm pilot study of a new smartphone app to support adherence to PrEP medication for HIV prevention in public clinics in Virginia.

DETAILED DESCRIPTION:
Testing the impact of a smart phone application's impact on PrEP uptake and adherence.

The app features daily medication reminders, daily mood and stress evaluations, a community message board for social support, and patient-provider secure, HIPAA compliant private messaging between patients and clinic providers. Participants will be recruited from VDH clinics. We will evaluate the adherence and uptake rates of PrEP among study participants. Usage data will be collected from the application, and from participant surveys at 30 day, 3 month, and 6 month study timepoints. Surveys will include questionnaires on medication adherence, empathy of providers, experiences with the app, stigma and disclosure attitudes, and social support, along with mental health screening. The study will be analyzed as a prospective one arm study by comparing baseline to 3M and 6M surveys, along with examining and characterizing app usage across time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* one or considering being on PrEP for HIV prevention
* Patient at a VDH or VDH funded clinic
* ability to read at a 5th grade reading level

Exclusion Criteria:

* HIV positive individuals
* Persons under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Adherence | 6 months
  Overall percentage of PrEP medication adherence

SECONDARY OUTCOMES:
Usability | 6 months
  How usable is the app to both patient participants and provider participants

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Department of Health, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No